CLINICAL TRIAL: NCT05780671
Title: The Effectiveness of Supplemental Oxygen Therapy in Patients Receiving Acute Migraine Treatment in the Emergency Department
Brief Title: Oxygen in Migraine Treatment
Status: Completed | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, GÜLŞAH ÇIKRIKÇI IŞIK, Associated Proffesor, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: E-66175679-514.05.02-1015712
Record Dates: First submitted 2023-03-13; First posted 2023-03-22 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Migraine Headache; Oxygen
MeSH Terms: conditions — Migraine Disorders | interventions — Oxygen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oxygen receiving group: patients diagnosed as headcahe related to migraine without aura who received supplemental oxygen together with the standart theraphy
  Interventions: Other: oxygen
- standart group: patients diagnosed as headcahe related to migraine without aura who received standart theraphy only.

INTERVENTIONS:
Other: oxygen — inhaled oxygen 10L/min with face mask for 1 hour
  Groups: Oxygen receiving group

SUMMARY:
IIn this study, the investigators planned to investigate effectiveness of supplemental oxygen in patients (18-65 years) who were diagnosed as headache related to migraine without aura in the emergency department (ED).

Patients who will be ordered standard migraine therapy (50 mg dexketoprofen and 10 mg metoclopramide HCl in 100 cc normal saline IV) by the physician blind to research, will be evaluated by the researchers before the treatment and patients met the study criteria will be included. Included patients randomly divided to two group, study group will receive supplemental oxygen with face mask for 1 hour.

Patients' visual analog score (VAS) will be measured at 0th, 15th, 30th and 60th minute of treatment. If there will not be a 50% decrease at VAS score from the beginning, patients will be examined again by the physician again. Patients who will be ordered 100 mg tramadol as rescue therapy by the physician, will be continued to observed, VAS scores will be measured at 120th minute again.

To avoid drug related bias, patients who will be ordered any other drug for primary care or rescue treatment other than mentioned above will not be included into the study.

ELIGIBILITY:
Inclusion Criteria:

with their medical history and ED evaluation being diagnosed as migraine related headache according to HIS 2018 classification, having VAS >40 at the beginning of the treatment, accepting to participate patient group who received standard migraine therapy (50 mg dexketoprofen and 10 mg metoclopramide HCl in 100 cc normal saline iIV).

patient who received 100 mg tramadol as rescue therapy

Exclusion Criteria:

Taking any analgesic in 6 hours before admission, patients who were diagnosed with all other types of primary headaches (migraine with aura, migraine status, TTH, trigeminal autonomic cephalgia etc), patients using anticoagulants or have bleeding diathesis, pregnant and breastfeeding patients, patients had fever, patients diagnosed as secondary headaches, patients had focal neurologic findings, patients had heart, liver, or kidney failure, patients had peptic ulcer, patients had chronic obstructive pulmonary disease, patients had acute coronary syndrome, patients who were not stable hemodynamically patients who had history of acute dystonia or akathisia due to metoclopramide.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ED due to headache and who had a prior diagnosis of migraine without aura, were the candidates for study. Among those patients who had diagnosed as headache related to migraine without aura according to 2018 criteria of International Headache Society (IHS) with a visual analog scale (VAS) value above "40" at the 0th minute of treatment were included into the study.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
examine effect of oxygen therapy in pain management of acute migraine attacks in emergency department. | until December 2023
  comprasion of VAS scores

SECONDARY OUTCOMES:
Rate of pain relief and need for additional analgesics were determined as secondary outcomes to be evaluated. | until december 2023

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Ankara Ataturk Sanatorium TRH, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
all data and statistical analyzes